CLINICAL TRIAL: NCT07200674
Title: Interest of High-speed Centrifugation for Measuring Anti-Xa Activity on Lipemic Plasma
Acronym: LCGV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9241
Record Dates: First submitted 2025-03-26; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia; High-Speed Centrifugation; Anti-Xa Activity; Lipemic Plasma; Hemostasis; Hematology
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some hemostasis techniques require spectrophotometric measurements. These are then subject to interference from the sample's lipemia (postprandial, hypertriglyceridemia, etc.), which risks distorting the results; this is estimated to affect 0.5 to 2.5% of samples.

This is particularly the case for anti-Xa activity, a critical test used to monitor anticoagulant treatments.

To date, the HUS Hematology Laboratory does not have or is aware of any alternative method to overcome this interference, and is unable to perform anti-Xa activity when the sample has excessive lipemia. This study will evaluate, on samples from routine care artificially overloaded with lipids, the effectiveness of a high-speed centrifugation process (10,800g for 10 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Patient anticoagulated with an anti-Xa (UFH, LMWH, fondaparinux, danaparoid, apixaban, rivaroxaban)
* Sample sent to the HUS Hematology Laboratory and analyzed for measurement of the anti-Xa activity of an anticoagulant as part of routine care

Exclusion Criteria:

* Patient with a basal lipidemic sample
* Sample of insufficient volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years) anticoagulated with an anti-Xa
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
To determine whether high-speed centrifugation (10,800g for 10 minutes) effectively separates the lipid fraction from the rest of the plasma | Up to 10 minutes
  To determine whether high-speed centrifugation (10,800g for 10 minutes) effectively separates the lipid fraction from the rest of the plasma, in order to measure anti-Xa activity, and to ensure that this process does not interfere with this measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - Unité d'Hémostase - CHU de Strasbourg - France, Strasbourg, France